CLINICAL TRIAL: NCT00999206
Title: Randomized, Double-Blind Study to Assess Safety, Immunogenicity, and Lot Consistency of Solvay's Cell-Derived Influenza Vaccine and Its Non-Inferiority Compared to Influvac®.
Brief Title: Study Measuring the Safety, Immunogenicity and Lot Consistency of Cell Derived Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Biologicals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S203.3.013
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; CHMP criteria
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Biological: Influenza Vaccine
- 2 (Experimental)
  Interventions: Biological: Influenza Vaccine
- 3 (Experimental)
  Interventions: Biological: Influenza Vaccine
- 4 (Active Comparator)
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Vaccine — surface antigen, inactivated, prepared in cell cultures
  Arms: 3
Biological: Influenza Vaccine — surface antigen, inactivated, prepared in egg (influvac ®)
  Arms: 4
Biological: Influenza Vaccine — surface antigen, inactivated, prepared in cell cultures
  Arms: 1
Biological: Influenza Vaccine — surface antigen, inactivated, prepared in cell cultures
  Arms: 2

SUMMARY:
A phase 3 study to obtain additional safety and immunogenicity data on Solvay's cell-derived seasonal trivalent subunit influenza vaccine in adult and elderly subjects without significant illnesses and to demonstrate consistency of the immunogenicity of the three lots of the same vaccine, comparison of cell-derived vaccine to Solvay's egg-derived vaccine including assessment of non-inferior immunogenicity

ELIGIBILITY:
Inclusion Criteria

1. Female or male subjects >= 18 years of age (adults >= 18 to < =60 years of age or elderly >= 61 years of age).
2. Willing and able to give informed consent before any protocol procedures are performed.
3. Able to adhere to visit schedules and all protocol required study procedures.
4. Being in good health as determined by medical history, physical examination and clinical judgment of the investigator (subjects may have underlying illnesses such as hypertension, diabetes, ischemic heart disease or hypothyroidism, as long as the disease is well controlled. If on medication for a condition, the medication dose must have been stable for at least 3 months preceding study vaccination).

Exclusion Criteria

1. Influenza vaccination or laboratory confirmed influenza infection within six months preceding the date of study vaccination or planning an influenza vaccination during the three weeks after study vaccination (i.e. between study Day 1 and study Day 22).
2. Presence of any significant condition that may prohibit inclusion as determined by the Investigator.
3. A serious adverse reaction after a previous (influenza) vaccination.
4. A history of Guillain-Barré syndrome.
5. Known to be allergic to constituents of the study vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3138 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Anti-HA antibody titers and derived parameters seroprotection, seroconversion and fold increase | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hanka de Voogd, MD, Study Director — Abbott Healthcare Products B.V.
Locations (19):
- Australia (13):
  - Site Reference ID/Investigator# 44652, Adelaide
  - Site Reference ID/Investigator# 44662, Auchenflower
  - Site Reference ID/Investigator# 44651, Blacktown
  - Site Reference ID/Investigator# 44659, Blacktown
  - Site Reference ID/Investigator# 44647, Broadmeadow
  - Site Reference ID/Investigator# 44649, Caboolture
  - Site Reference ID/Investigator# 44646, Carina Heights
  - Site Reference ID/Investigator# 44650, Herston
  - Site Reference ID/Investigator# 44663, Hornsby
  - Site Reference ID/Investigator# 44645, Kippa-Ring
  - Site Reference ID/Investigator# 44644, Malvern East
  - Site Reference ID/Investigator# 44648, Maroubra Junction
  - Site Reference ID/Investigator# 44643, Sherwood
- New Zealand (6):
  - Site Reference ID/Investigator# 44653, Christchurch
  - Site Reference ID/Investigator# 44658, Dunedin
  - Site Reference ID/Investigator# 44656, Grafton
  - Site Reference ID/Investigator# 44655, Rotorua
  - Site Reference ID/Investigator# 44654, Tauranga
  - Site Reference ID/Investigator# 44657, Wellington